CLINICAL TRIAL: NCT04623008
Title: Using Mental Imagination to Prevent Excessive Gestational Weight Gain in Overweight and Obese Pregnant Women
Acronym: MAWI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Mei-Wei Chang, Assoicate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019H0441
Record Dates: First submitted 2020-10-19; First posted 2020-11-10 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Obesity; Weight Gain, Maternal
Keywords: pregnant women; intervention
MeSH Terms: conditions — Obesity; Gestational Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal-Oriented Episodic Future Thinking (GOEFT) Intervention (Experimental): In addition to usual prenatal care, intervention participants will receive a 20-week intervention via web and individual health counseling. The intervention topics focus on stress management, healthy eating, and physical activity.
  Interventions: Behavioral: Goal-Oriented Episodic Future Thinking
- Usual Prenatal Care (No Intervention): The usual prenatal care group will receive usual care from their providers

INTERVENTIONS:
Behavioral: Goal-Oriented Episodic Future Thinking — Individuals in the intervention group will receive a 20-week web-based intervention and individual health coaching focused on stress management, healthy eating and physical activity.
  Arms: Goal-Oriented Episodic Future Thinking (GOEFT) Intervention

SUMMARY:
Moms Are Worth It is a lifestyle behavior intervention study aims to prevent excessive gestational weight gain in overweight or obese pregnant women through promotion of the stress management, healthy eating, and physical activity. Eligible women will be randomly assigned to a usual care or an intervention plus usual care group. The intervention will last 20 weeks and will be delivered via weekly web and individual health coaching session (10 of them)

DETAILED DESCRIPTION:
Current effective lifestyle behavior intervention studies aimed to prevent excessive gestational weight gain (EGWG) in overweight or obese pregnant women have limited practicality, scalability, and sustainability because of high participant burden and excessive cost for clinical practice. Also, prior studies paid little or no attention to motivation, emotion and cognition, all of which are critical to motivate and enable individuals to engage in healthy lifestyle behaviors and achieve positive health outcomes. A promising approach to prevent EGWG in overweight or obese pregnant women is through goal-oriented episodic future thinking (GOEFT). This pilot randomized controlled trial, aims to prevent EGWG in overweight or obese pregnant women. The proposed self-directed, web-based GOEFT intervention will focus on increasing motivation (autonomous motivation and self-efficacy) and improving emotion (emotion control and stress) and cognition (executive function, ExF), thus promoting healthy lifestyle behaviors. This will lead to prevention of EGWG and a reduced rate of gestational diabetes, gestational hypertension, cesarean delivery and fetal macrosomia. Our intervention will last 20 weeks (starting at 17 week-gestation). Participants (N = 90; 50% White, 50% minority) will be recruited and enrolled from prenatal care clinics at The Ohio State University Wexner Medical Center and be randomly assigned to our GOEFT intervention (n = 45) or usual care (n = 45). All participants will be assessed at baseline (<17 week-gestation, T1), 24-27 week-gestation (T2) and 35-37 week-gestation (T3). Specific aims are (1) to determine feasibility of the GOEFT intervention: recruitment, randomization, retention and intervention implementation, (2) to investigate the potential efficacy of the intervention on gestational weight gain and maternal and birth outcomes, (3) to investigate the potential impact of the intervention on lifestyle behaviors and (4) to investigate the potential impact of the intervention on motivation, emotion and cognition.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be pregnant women ≤ 13 week-gestation with a single fetus as assessed by ultrasound.
* Participants must also have self-reported pre-pregnancy body mass index (BMI) of 25.0-45.0 kg/m2 and height (height and weight to compute body mass index).
* Ability to read and speak English,
* Age of 18-45 years,
* Access to a working smart phone with unlimited text messaging,
* Access to internet,
* Receipt of prenatal care from our collaborating clinics and plan to deliver the baby at The Ohio State University (OSU) Wexner Medical Center,
* Resident of Franklin Count,
* Committed to the 20-week intervention.

Exclusion Criteria:

* Self-reported history of ≥ 3 miscarriages,
* Planned termination of the pregnancy,
* Diagnosed hypertension and/or type 1 or 2 diabetes,
* History of or current diagnosis of an eating disorder,
* Serious current physical disease (e.g., renal disease or cancer),
* Past bariatric surgery,
* Current or history of substance abuse in the past 6 months,
* Current treatment for a serious psychological disorder (e.g., schizophrenia and bipolar disorder),
* Contraindications to walking,
* Consented women will become not eligible to participate in the study if they are not randomized by 16-week 6 days gestation. This is because the study intervention starts ≤ 17 weeks gestation.
* Women will become not ineligible for participation if they did not complete the baseline data.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants need to be pregnant women.
Enrollment: 70 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Wei Chang, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February, 2021 and March, 2022, Clinicians at collaborating sites referred pregnant patients to our study. The study research assistants screened the potential participants for eligibility over the phone.
Pre-assignment Details: Eligible participants completed baseline measures; had body mass index (BMI) of 25.0-45.0 kg/m2 (calculated using self reported height and pre-pregnancy weight) and be between 18 and 45 years old. We excluded potential participants with self-reported history of ≥ 3 miscarriages, eating disorder, and diagnosed hypertension and type 1 or 2 diabetes, or contraindications to walking.
Period: Baseline to T2
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Started | 35 | 35
Completed | 31 | 33
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 4 | 2
Period: Baseline to T3
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Started (This Timepoint measures from Baseline to T3 (the full timeframe of the study). The study measured from Baseline to each individual data collection period, in addition to the midpoint to the end. Therefore all 70 participants started this Timepoint.) | 35 | 35
Completed | 31 | 33
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 4 | 2
Period: T2 toT3
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Started | 31 | 33
Completed | 31 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (4.3) | 32.0 (3.8) | 32.2 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic White | 0 | 3 | 3
  Asian | 1 | 2 | 3
  Non-Hispanic Black | 8 | 2 | 10
  Non-Hispanic White | 25 | 26 | 51
  More than one race | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70
Marital Status [Count of Participants; unit: Participants]
  Single, never married | 3 | 3 | 6
  Married | 31 | 32 | 63
  In a domestic partnership | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Body Weight
Description: Data extracted from electronic medical record
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 24-27 week-gestation (T2)
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 31 | 33
percentage change | 10.9 (8.8) | 9.6 (11.0)

2. Primary Outcome: Percent Change in Body Weight
Description: Data extracted from electronic medical record
Time Frame: 24-27 week-gestation (T2) to 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 31 | 33
percent change | 14.0 (7.1) | 13.9 (12.6)

3. Primary Outcome: Percent Change in Body Weight
Description: Data extracted from electronic medical record
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 31 | 33
percent change | 24.9 (12.2) | 23.5 (10.8)

4. Secondary Outcome: Percentage of Participants Diagnosed With Gestational Diabetes
Description: Data extracted from electronic medical record. Percentage of participants who were diagnosed with Gestational Diabetes during the study timeframe.
Time Frame: 24-27 week-gestation (T2) to 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 31 | 33
percentage of participants | 4 (12.9) | 5 (15.2)

5. Secondary Outcome: Percentage of Participants Diagnosed With Gestational Hypertension
Description: Data extracted from electronic medical record. Percentage of participants diagnosed with Gestational Hypertension in the study timeframe.
Time Frame: 24-27 week-gestation (T2) to 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: percent of participants
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 31 | 33
percent of participants | 4 (12.9) | 2 (6.1)

6. Secondary Outcome: Percentage of Participants With Cesarean Delivery
Description: Data extracted from electronic medical record. Percentage of participants who experienced Cesarean Delivery.
Time Frame: 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 31 | 33
percentage of participants | 9 (29.0) | 9 (27.3)

7. Secondary Outcome: Newborn Body Weight
Description: Data extracted from electronic medical record. Newborn Body Weight taken at birth.
Time Frame: 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 31 | 33
grams | 3493 (327.7) | 3503 (483.2)

8. Secondary Outcome: Percentage of Participants With Premature (<37 Weeks Gestation) Births
Description: Gestational age for each participant was extracted from electronic medical record and births before 37 weeks gestation were considered to be premature. The number of premature births was averaged within the study groups.
Time Frame: 35-37 week-gestation (T3)
Measure: Count of Participants; unit: Participants
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 31 | 33
Participants | 0 | 3

9. Secondary Outcome: Percentage of Change in Dietary Intake Behaviors - Caloric Intake (Kcal)
Description: Assessed using the National Cancer Institute Automated Self-Administered 24-hour Recall (ASA24). Participants completed 24-hour Dietary Recalls on two random days over a week. The variable of interest - calories (Kcal) - values for the 2 24-hour periods were added to ascertain the total amount consumed at the specific data collection time periods.
  Data from Baseline (T1) was compared to that collected at T2 for each participant and averaged for an aggregate score. Positive numbers represent an increase in calories consumed, negative numbers represent a decrease in calories consumed.
  Only participants who completed 2 days worth of dietary data were included in this analysis.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 24-27 week-gestation (T2)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 12 | 24
percentage of change | 162.9 (545.7) | -149 (655.9)

10. Secondary Outcome: Percentage of Change in Dietary Intake Behaviors - Fat (gm)
Description: Assessed using the National Cancer Institute Automated Self-Administered 24-hour Recall (ASA24). Participants completed 24-hour Dietary Recalls on two random days over a week. The variable of interest - fat (gm) - values for the 2 24-hour periods were added to ascertain the total amount consumed at the specific data collection time periods.
  Data from Baseline (T1) was compared to that collected at T2 for each participant and averaged for an aggregate score. Positive numbers represent an increase in fat consumed, negative numbers represent a decrease in fat consumed.
  Only participants who completed 2 days worth of dietary data were included in this analysis.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 24-27 week-gestation (T2)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 12 | 24
percentage of change | 9.89 (32.74) | -0.84 (40.73)

11. Secondary Outcome: Percentage of Change in Dietary Intake Behaviors - Fruit (Cup)
Description: Assessed using the National Cancer Institute Automated Self-Administered 24-hour Recall (ASA24). Participants completed 24-hour Dietary Recalls on two random days over a week. The variable of interest - fruit (cup) - values for the 2 24-hour periods were added to ascertain the total amount consumed at the specific data collection time periods.
  Data from Baseline (T1) was compared to that collected at T2 for each participant and averaged for an aggregate score. Positive numbers represent an increase in fruit consumed, negative numbers represent a decrease in fruit consumed.
  Only participants who completed 2 days worth of dietary data were included in this analysis.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 24-27 week-gestation (T2)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 12 | 24
percentage of change | 0.63 (2.50) | -0.25 (1.37)

12. Secondary Outcome: Percentage of Change in Dietary Intake Behaviors - Vegetable (Cup)
Description: Assessed using the National Cancer Institute Automated Self-Administered 24-hour Recall (ASA24). Participants completed 24-hour Dietary Recalls on two random days over a week. The variable of interest - vegetables (cup) - values for the 2 24-hour periods were added to ascertain the total amount consumed at the specific data collection time periods.
  Data from Baseline (T1) was compared to that collected at T2 for each participant and averaged for an aggregate score. Positive numbers represent an increase in vegetables consumed, negative numbers represent a decrease in vegetables consumed.
  Only participants who completed 2 days worth of dietary data were included in this analysis.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 24-27 week-gestation (T2)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 12 | 24
percentage of change | 0.18 (1.65) | 0.22 (0.84)

13. Secondary Outcome: Percentage of Change in Dietary Intake Behaviors - Added Sugars (Teaspoon or 4gm)
Description: Assessed using the National Cancer Institute Automated Self-Administered 24-hour Recall (ASA24). Participants completed 24-hour Dietary Recalls on two random days over a week. The variable of interest - added sugars teaspoon or 4 gm) - values for the 2 24-hour periods were added to ascertain the total amount consumed at the specific data collection time periods.
  Data from Baseline (T1) was compared to that collected at T2 for each participant and averaged for an aggregate score. Positive numbers represent an increase in added sugars consumed, negative numbers represent a decrease in added sugars consumed.
  Only participants who completed 2 days worth of dietary data were included in this analysis.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 24-27 week-gestation (T2)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 12 | 24
percentage of change | 2.35 (7.26) | -2.99 (8.16)

14. Secondary Outcome: Percentage of Change in Dietary Intake Behaviors - Caloric Intake (Kcal)
Description: Assessed using the National Cancer Institute Automated Self-Administered 24-hour Recall (ASA24). Participants completed 24-hour Dietary Recalls on two random days over a week. The variable of interest - calories (Kcal) - values for the 2 24-hour periods were added to ascertain the total amount consumed at the specific data collection time periods.
  Data from Baseline (T1) was compared to that collected at T3 for each participant and averaged for an aggregate score. Positive numbers represent an increase in calories consumed, negative numbers represent a decrease in calories consumed.
  Only participants who completed 2 days worth of dietary data were included in this analysis.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 15 | 18
percentage of change | 98.34 (651.4) | -217 (627.0)

15. Secondary Outcome: Percentage of Change in Dietary Intake Behaviors - Fat Intake (gm)
Description: Assessed using the National Cancer Institute Automated Self-Administered 24-hour Recall (ASA24). Participants completed 24-hour Dietary Recalls on two random days over a week. The variable of interest - fat (gm) - values for the 2 24-hour periods were added to ascertain the total amount consumed at the specific data collection time periods.
  Data from Baseline (T1) was compared to that collected at T3 for each participant and averaged for an aggregate score. Positive numbers represent an increase in fat consumed, negative numbers represent a decrease in fat consumed.
  Only participants who completed 2 days worth of dietary data were included in this analysis.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 15 | 18
percentage of change | 15.18 (43.30) | -11.1 (38.83)

16. Secondary Outcome: Percentage of Change in Dietary Intake Behaviors - Fruit Intake (Cups)
Description: Assessed using the National Cancer Institute Automated Self-Administered 24-hour Recall (ASA24). Participants completed 24-hour Dietary Recalls on two random days over a week. The variable of interest - fruit (cup) - values for the 2 24-hour periods were added to ascertain the total amount consumed at the specific data collection time periods.
  Data from Baseline (T1) was compared to that collected at T3 for each participant and averaged for an aggregate score. Positive numbers represent an increase in fruit consumed, negative numbers represent a decrease in fruit consumed.
  Only participants who completed 2 days worth of dietary data were included in this analysis.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 15 | 18
percentage of change | 0.12 (1.07) | 0.19 (1.32)

17. Secondary Outcome: Percentage of Change in Dietary Intake Behaviors - Vegetable Intake (Cups)
Description: Assessed using the National Cancer Institute Automated Self-Administered 24-hour Recall (ASA24). Participants completed 24-hour Dietary Recalls on two random days over a week. The variable of interest - vegetable (cup) - values for the 2 24-hour periods were added to ascertain the total amount consumed at the specific data collection time periods.
  Data from Baseline (T1) was compared to that collected at T3 for each participant and averaged for an aggregate score. Positive numbers represent an increase in vegetables consumed, negative numbers represent a decrease in vegetables consumed.
  Only participants who completed 2 days worth of dietary data were included in this analysis.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 15 | 18
percentage of change | -0.11 (1.65) | 0.08 (1.34)

18. Secondary Outcome: Percentage of Change in Dietary Intake Behaviors - Added Sugars Intake (gm)
Description: Assessed using the National Cancer Institute Automated Self-Administered 24-hour Recall (ASA24). Participants completed 24-hour Dietary Recalls on two random days over a week. The variable of interest - added sugars (teaspoon or 4 gm) - values for the 2 24-hour periods were added to ascertain the total amount consumed at the specific data collection time periods.
  Data from Baseline (T1) was compared to that collected at T3 for each participant and averaged for an aggregate score. Positive numbers represent an increase in added sugars consumed, negative numbers represent a decrease in added sugars consumed.
  Only participants who completed 2 days worth of dietary data were included in this analysis.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 15 | 18
percentage of change | 3.08 (13.27) | -2.28 (10.96)

19. Secondary Outcome: Percentage of Change in Physical Activity - 7-Day Metabolic Equivalent of Task (MET)
Description: Assessed using Actigraph (GT3x), an objective measurement of physical activity. Investigators distributed the Actigraph in person participants' home (T2 and T3) to wear at the wrist at least seven consecutive days (≥ 10 hours/per day).
  The variable of interest - 7-day MET - values for the period was added to ascertain the total amount at the specific data collection time periods.
  Data from Baseline (T1) was compared to that collected at T2 for each participant and averaged for an aggregate score. Positive numbers represent an increase in physical activity negative numbers represent a decrease in physical.
  Only participants who completed the minimum requirement for reporting [wear at the wrist at least seven consecutive days (≥ 10 hours/per day)] were included in the analysis.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 24-27 week-gestation (T2)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 23 | 30
percentage of change | 1.77 (9.31) | 3.65 (9.85)

20. Secondary Outcome: Percentage of Change in Physical Activity - 7-Day Metabolic Equivalent of Task (MET)
Description: Assessed using Actigraph (GT3x), an objective measurement of physical activity. Investigators distributed the Actigraph in person participants' home (T2 and T3) to wear at the wrist at least seven consecutive days (≥ 10 hours/per day).
  The variable of interest - 7-day MET - values for the period was added to ascertain the total amount at the specific data collection time periods.
  Data from Baseline (T1) was compared to that collected at T3 for each participant and averaged for an aggregate score. Positive numbers represent an increase in physical activity negative numbers represent a decrease in physical.
  Only participants who completed the minimum requirement for reporting [wear at the wr
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 18 | 28
percentage of change | 3.06 (7.09) | 1.13 (11.40)

21. Secondary Outcome: Change in Autonomous Motivation for Physical Activity
Description: Will be measured using Treatment Self-Regulation Questionnaire (6 items) to measure autonomous motivation for Physical Activity (6 items)
  Values are: 1 - Not At All True, 2, 3, 4 - Somewhat True, 5, 6, 7 - Very True
  The investigators will sum 6 items to create a composite score, ranging from 6 to 42.
  Higher scores indicate higher autonomous motivation for Physical Activity.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 24-27 week-gestation (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 11 | 26
score on a scale | 1.64 (2.80) | 0.92 (5.55)

22. Secondary Outcome: Change in Autonomous Motivation for Physical Activity
Description: as for outcome 21
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 14 | 18
score on a scale | -1.60 (4.79) | -1.26 (6.81)

23. Secondary Outcome: Change in Autonomous Motivation for Stress Management
Description: Will be measured using Treatment Self-Regulation Questionnaire (6 items) to measure autonomous motivation for stress management (6 items)
  Values are: 1 - Not At All True, 2, 3, 4 - Somewhat True, 5, 6, 7 - Very True
  The investigators will sum 6 items to create a composite score, ranging from 6 to 42.
  Higher scores indicate higher autonomous motivation for stress management.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 24-27 week-gestation (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 11 | 26
score on a scale | -0.09 (2.84) | 1.54 (4.96)

24. Secondary Outcome: Change in Autonomous Motivation for Stress Management
Description: Will be measured using Treatment Self-Regulation Questionnaire (6 items) to measure autonomous motivation for stress management (6 items)
  Values are: 1 - Not At AllTrue, 2, 3, 4 - Somewhat True, 5, 6, 7 - Very True
  The investigators will sum 6 items to create a composite score, ranging from 6 to 42.
  Higher scores indicate higher autonomous motivation for stress managment.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 14 | 18
score on a scale | -0.27 (5.38) | -0.68 (6.71)

25. Secondary Outcome: Change in Autonomous Motivation for Healthy Eating
Description: Will be measured using Treatment Self-Regulation Questionnaire (6 items) to measure autonomous motivation for Healthy Eating (6 items)
  Values are: 1 - Not At All True, 2, 3, 4 - Somewhat True, 5, 6, 7 - Very True
  The investigators will sum 6 items to create a composite score, ranging from 6 to 42.
  Higher scores indicate higher autonomous motivation for Healthy Eating.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 24-27 week-gestation (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 11 | 26
score on a scale | 2.00 (3.29) | 0.38 (4.53)

26. Secondary Outcome: Change in Autonomous Motivation for Healthy Eating
Description: as for outcome 25
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 14 | 18
score on a scale | -0.93 (5.75) | -2.95 (6.70)

27. Secondary Outcome: Change in Healthy Eating Self-efficacy
Description: Will be measured using a "Survey for Healthy Eating Self-efficacy" (8 items)
  Values are: 1 - Not At All Confident, 2 - Not Too Confident, 3 - Somewhat Confident, 4 - Very Confident.
  The investigators will sum all 8 items to create a composite score, ranging from 8 to 32.
  The higher score, the higher healthy eating self-efficacy.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 24-27 week-gestation (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 11 | 26
score on a scale | 2.27 (3.58) | 1.31 (3.58)

28. Secondary Outcome: Change in Healthy Eating Self-efficacy
Description: Will be measured using a "Survey for Healthy Eating Self-efficacy" (8 items)
  Values are: 1 - Not At All Confident, 2 - Not Too Confident, 3 - Somewhat Confident, 4 - Very Confident
  The investigators will sum all 8 items to create a composite score, ranging from 8 to 32. The higher score, the higher healthy eating self-efficacy.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 14 | 18
score on a scale | 2.80 (3.32) | 0.84 (4.45)

29. Secondary Outcome: Change in Coping Self-efficacy
Description: Will be measured using a "Survey for Coping Self-efficacy" (10 items)
  Values are: 1 - Not At All Confident, 2 - Not Too Confident, 3 - Somewhat Confident, 4 - Very Confident
  The investigators will sum 10 items to create a composite score, ranging from 10 to 40.
  Higher scores indicate higher coping self-efficacy.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 24-27 week-gestation (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 11 | 26
score on a scale | 1.09 (4.72) | 1.35 (4.34)

30. Secondary Outcome: Change in Coping Self-efficacy
Description: as for outcome 29
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 14 | 18
score on a scale | 4.07 (6.06) | 1.21 (3.28)

31. Secondary Outcome: Change in Physical Activity Self-efficacy
Description: Will be measured using a "Survey for Physical Activity Self-efficacy" (10 items) that ask participants' confidence in performing the specific activity.
  Values are: 1 - Not At All Confident, 2 - Not Too Confident, 3 - Somewhat Confident, 4 - Very Confident
  The investigators will sum all 10 items to create a composite score, ranging from 10 to 40. The higher score, the higher physical activity self-efficacy.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 24-27 week-gestation (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 11 | 26
score on a scale | 2.45 (5.89) | 1.19 (4.42)

32. Secondary Outcome: Change in Physical Activity Self-efficacy
Description: as for outcome 31
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 14 | 18
score on a scale | 1.40 (5.17) | 2.00 (3.87)

33. Secondary Outcome: Change in Emotion Regulation
Description: The Emotion Regulation Questionnaire (10 items) was used to measure emotional control. The questionnaire asked participants to report the use of emotional regulatory process using a 7-point scale ranging from 1 (strongly disagree) to 7 (strongly agree). After revise coding 4 items, we summed responses of 10 items to create an emotional control score (ranged from 10 to 70). Higher scores indicated better emotional control.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 24-27 week-gestation (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 11 | 26
score on a scale | 3.64 (6.52) | -0.50 (5.26)

34. Secondary Outcome: Change in Emotion Regulation
Description: as for outcome 33
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 14 | 18
score on a scale | 2.73 (5.76) | -1.53 (6.26)

35. Secondary Outcome: Change in Perceived Stress
Description: Will be measured using The Perceived Stress Scale (10 items) that measures the degree to which situations in one's life are appraised as stressful.
  Values are: 0 - Never, 1 - Almost Never, 2 - Sometimes, 3 - Fairly Often, 4 - Very Often
  The investigators will sum 10 items to create a composite score, ranging from 0 to 40.
  The higher score, the higher levels of perceived stress.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 24-27 week-gestation (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 11 | 26
score on a scale | 1.73 (6.12) | 2.04 (5.39)

36. Secondary Outcome: Change in Perceived Stress
Description: as for outcome 35
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 14 | 18
score on a scale | -1.60 (6.23) | 0.72 (4.52)

37. Secondary Outcome: Change in Executive Function - Behavior Regulation
Description: The Behavior Rating Inventory of Executive Function-Adults (75 items) was used to measure executive function. This survey asked participants to rate self-regulation behaviors in the everyday environment using a 3-point Likert scale ranging from 0 (never) to 2 (often). This survey covers 2 main domains: behavior regulation (30 items) and metacognition (45 items). We summed responses to the 30 behavior regulation items to create a behavior regulation score. Behavior regulation scores range from 0-60. We used the same approach to create a composite score for metacognition. Higher scores indicated worse behavior regulation or metacognition. The scores from T1 were compared to scores for T2 to evaluate the effect of the intervention.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 24-27 week-gestation (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 11 | 26
score on a scale | 0.36 (5.71) | 1.88 (7.39)

38. Secondary Outcome: Change in Executive Function - Behavioral Regulation
Description: The Behavior Rating Inventory of Executive Function-Adults (75 items) was used to measure executive function. This survey asked participants to rate self-regulation behaviors in the everyday environment using a 3-point Likert scale ranging from 0 (never) to 2 (often). This survey covers 2 main domains: behavior regulation (30 items) and metacognition (45 items). We summed responses to the 30 behavior regulation items to create a behavior regulation score. Behavior regulation scores range from 0-60. We used the same approach to create a composite score for metacognition. Higher scores indicated worse behavior regulation or metacognition. The scores from T1 were compared to scores for T3 to evaluate the effect of the intervention.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 14 | 18
score on a scale | -0.43 (3.99) | -0.17 (5.22)

39. Secondary Outcome: Change in Executive Function - Metacognition
Description: The Behavior Rating Inventory of Executive Function-Adults (75 items) was used to measure executive function [31]. This survey asked participants to rate self-regulation behaviors in the everyday environment using a 3-point scale ranging from 0 (never) to 2 (often). This survey covers 2 main domains: behavior regulation (30 items) and metacognition (45 items). We summed responses to the 30 behavior regulation items to create a behavior regulation score. We used the same approach to create a composite score for metacognition. Metacognition scores range from 0-90. Higher scores indicated worse metacognition. The scores from T1 were compared to scores from T2 to evaluate the effect of the intervention.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 24-27 week-gestation (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 11 | 26
score on a scale | -8.36 (15.81) | 1.46 (12.21)

40. Secondary Outcome: Change in Executive Function - Metacognition
Description: The Behavior Rating Inventory of Executive Function-Adults (75 items) was used to measure executive function [31]. This survey asked participants to rate self-regulation behaviors in the everyday environment using a 3-point scale ranging from 0 (never) to 2 (often). This survey covers 2 main domains: behavior regulation (30 items) and metacognition (45 items). We summed responses to the 30 behavior regulation items to create a behavior regulation score. We used the same approach to create a composite score for metacognition. Metacognition scores range from 0-90. Higher scores indicated worse metacognition. The scores from T1 were compared to scores from T3 to evaluate the effect of the intervention.
Time Frame: Baseline: less than or equal to 16 week-gestation (T1) to 35-37 week-gestation (T3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
Number analyzed (Participants) | 14 | 18
score on a scale | -5.86 (11.37) | -1.78 (1.28)

ADVERSE EVENTS:
Time Frame: 20 Week period of study
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
  Additional criteria for Serious Adverse event was loss of pregnancy
Arm/Group | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention | Usual Prenatal Care
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 1/35 | 2/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Goal-Oriented Episodic Future Thinking (GOEFT) Intervention (N=35) | Usual Prenatal Care (N=35)
Loss of Pregancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT04623008/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT04623008/ICF_001.pdf